CLINICAL TRIAL: NCT06955273
Title: Multi-Centre Based Study Recognition of Atrial Fibrillation With the Corsano CardioWatch 287-2 System
Acronym: COR-AF
Status: Not yet recruiting | Type: Observational
Sponsor: Corsano Health B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: COR-AF
Record Dates: First submitted 2025-04-09; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF); Paroxysmal Atrial Fibrillation (PAF)
Keywords: wristband; wearable; atrial fibrillation; holter; ecg; remote monitoring; validation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Group A: patients receiving 24-48 hour holter monitoring as standard of care: Holter monitoring will be compared to continuous monitoring by the Corsano CardioWatch 287-2 across 24-48 hours to assess whether the amount and duration of AF episodes detected by the investigational device correspond to an ECG-holter reference across various demographic groups. Detection of atrial fibrillation with the Corsano CardioWatch 287-2 is done by optical photoplethysmography (PPG), after which atrial fibrillation can be confirmed with a 30-second ECG measurement. Additionally, all participants will be asked to perform 10 single-lead ECG's with the investigational device at standard timepoints (every 2 hours when awake), and when AF is detected (minimal 30 minutes time difference between alerts) across the 24-48 hours.
  Interventions: Device: Corsano CardioWatch 287-2
- Group B: patients diagnosed with (paroxysmal) AF presenting to the clinic for routine follow-up: Patients with a known diagnosis of (paroxysmal) atrial fibrillation presenting to the clinic for routine follow-up evaluation will be asked to eligibly participate in ECG-holter monitoring as well as continuous monitoring by the Corsano CardioWatch 287-2 across 24-48 hours. Similar to group A, these patients will also be asked to perform manual ECG measurements with the investigational device. Group B was added to ensure that a considerable amount of the included data includes periods with atrial fibrillation. As the results of a prior study (RECAMO study NCT05899959) show that the amount of patients in Group A with periods of atrial fibrillation is limited (7.0%).
  Interventions: Device: Corsano CardioWatch 287-2
- Group C: patients diagnosed with (paroxysmal) AF registered in a patient organisation: Patients with a known diagnosis of (paroxysmal) atrial fibrillation registered in a patient organisation for patients with AF will be asked to eligibly participate in ECG-holter monitoring as well as continuous monitoring by the Corsano CardioWatch 287-2 across 24-48 hours. Similar to group A and B, these patients will also be asked to perform manual ECG measurements with the investigational device. For this group two (virtual) visits will be scheduled before (visit a) and after (visit b) the study period. In visit a) additional information regarding the study will be provided and potential alarm signals will be screened to ensure the patient does not participate in the trial in case direct medical attention is required. If the patient does not show any alarm signals they will be asked to provide informed consent. Once informed consent is provided all materials will be mailed to them via postal services after which they can perform the measurements and return the materials via postal
  Interventions: Device: Corsano CardioWatch 287-2
- Group D: patients receiving a 12-lead ECG at the outpatient clinic as standard of care.: Participants in this group will wear the CardioWatch 287-2 during the standard 12-lead ECG recordings conducted in the outpatient clinic. Patients will be asked to perform a manual ECG spot-check with the investigational device during (if not feasible directly before), and immediately following the 12-lead ECG. Furthermore, the CardioWatch 287-2 will be worn for at least 5 minutes prior to and following the 12-lead ECG. Although these recordings are brief, this group was included to enhance the study population's size and demographic diversity while minimizing the burden on both patients and hospital staff. This group is expected to consist of both non-AF and AF patients, providing valuable insights into the investigational device's performance in a setting similar to its intended real-world application.
  Interventions: Device: Corsano CardioWatch 287-2

INTERVENTIONS:
Device: Corsano CardioWatch 287-2 — Patients receive monitoring of their heart rhythm by the CardioWatch 287-2 next to monitoring of their heart rhythm by either a 24-48 holter or a short in-clinic 12-lead ECG monitoring.

SUMMARY:
This concerns a multi-center, single-arm, diagnostic accuracy study. In this study, a wristband that monitors heart rythm is assessed in clinical and free living conditions. The performance of the wristband in detecting atrial fibrillation and normal sinus rhythms will be compared to a short 12-lead ECG or 24-hour holter.

To ensure that both patients with and without atrial fibrillation are included whilst limiting the burden on patients and hospital staff, four groups of patients are being recruited:

* Group A: patients receiving an ECG holter at the outpatient clinic for 24-48 hours of remote monitoring
* Group B: patients diagnosed with (paroxysmal) AF presenting to the clinic for routine follow-up evaluation.
* Group C: patients diagnosed with (paroxysmal) AF registered in a patient organisation for patients with AF.
* Group D: patients receiving a 12-lead ECG at the outpatient clinic as standard of care.

The secondary outcomes of the study focus on assessing the primary outcomes in light of demographic subgroups, patient physical activity and the signal quality index.

DETAILED DESCRIPTION:
Rationale:

Wearables have the potential to monitor patients remotely. The Corsano CardioWatch 287-2 is such a medical device that can monitor atrial fibrillation. The device has been validated using clinical trials in hospitals, but evaluation in the intended remote setting across various demographic groups is lacking.

Primary objective:

To compare episodes of atrial fibrillation across 30-second intervals detected by the Corsano CardioWatch 287-2 with episodes of atrial fibrillation detected by conventional Holter monitoring across 24-48 hours or short in-clinic 12-lead ECG based on the positive predictive value, negative predictive value, sensitivity and specificity.

Secondary objective: To compare the number of atrial fibrillation episodes greater than 6 minutes, 1 hour, 6 hours, and 12 hours duration detected by the CardioWatch 287-2 and with the number of these specific episodes detected by conventional Holter across 24-48 hours days. As well as to assess primary outcomes in light of demographic subgroups, patient activity and the signal quality index.

Study population:

One group (A) receiving an ECG monitoring holter for the duration of 24-48 hours days as part of standard care for atrial fibrillation screening. Besides, one group (B) diagnosed with (paroxysmal) without indication for holter monitoring according to standard of care AF presenting to the clinic for routine follow-up evaluation. Adding, one group (C) diagnosed with (paroxysmal) and registered in a patient organisation for patients with AF. Finally, one group (D) receiving in-clinic 12-lead ECG monitoring as part of standard of care.

Study design:

This concerns a multi-center, single-arm, diagnostic accuracy study.

Four different groups of patients will be approached for participation in the trial:

* Group A: patients receiving an ECG holter at the outpatient clinic for 24-48 hours of remote monitoring
* Group B: patients diagnosed with (paroxysmal) AF presenting to the clinic for routine follow-up evaluation.
* Group C: patients diagnosed with (paroxysmal) AF registered in a patient organisation for patients with AF.
* Group D: patients receiving a 12-lead ECG at the outpatient clinic as standard of care.

Groups A, B and C will receive ECG holter monitoring as well as continuous monitoring by the Corsano CardioWatch 287-2 across 24-48 hours to assess whether the amount and duration of AF episodes detected by the investigational device correspond to the gold standard. Detection of atrial fibrillation with the Corsano CardioWatch 287-2 is done by optical photoplethysmography (PPG), after which atrial fibrillation can be confirmed with a 30-second ECG measurement. Additionally, all participants will be asked to perform 10 single-lead ECG's at standard timepoints (approx. every 2 hours when awake) across the 24-48 hours as well as additional ECG measurements in case of AF (at least 30 minutes between alerts). Group B was added to ensure that a considerable amount of the included data includes periods with atrial fibrillation. As the results of a prior study (RECAMO study NL NL83281.000.22) show that the amount of patients in Group A with periods of atrial fibrillation is limited (7.0%). Furthermore, Group C was added to limit the additional workload for hospital staff and ensure inclusion of a diverse patient population from different demographic and ethnical groups. For this group two (virtual) visits will be scheduled before and after the study period to detect any alarming signals before participation in the study and to share and explain the results after study completion. Finally, group D, a group receiving a short in-clinic 12-lead ECG as standard of care was added to ensure the inclusion of a broad and sizable demographic group whilst keeping the burden on the patient and hospital staff limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms indicative of cardiac arrhythmias receiving 24-48 hour ECG holter for home monitoring or in-clinic 12-lead ECG per doctor prescription OR previous diagnosis of arrhythmia presenting to the clinic for routine follow-up evaluation
* Age ≥ 22 years old
* Able to provide informed consent.
* Proficient in written and spoken Dutch or English, defined by self-report of comfort reading, writing, and speaking Dutch or English.

Exclusion Criteria:

* Clinical conditions that in the opinion of the Investigator would compromise the safety of the patient or ability to complete the protocol;
* Unable to wear the Corsano CardioWatch 287 due to reasons such as allergic reactions, wounds, amputations etc.;
* Unable or not willing to receive ECG monitoring;
* Unable or not willing to sign informed consent;

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population for groups A-B-D includes patients visiting the outpatient clinic of at least 4 different hospitals, of which one is located in the Netherlands (Reinier de Graaf Gasthuis, Delft) and three are located in different locations across the USA.
  GROUP A Patients receiving an ECG holter at the outpatient clinic for 24 hours of remote monitoring (standard of care)
  GROUP B Patients diagnosed with (paroxysmal) AF presenting to the clinic for routine follow-up evaluation (NOT necessarily standard of care)
  GROUP C Patients diagnosed with (paroxysmal) AF registered in a patient organisation for patients with AF (standard of care)
  GROUP D Patients receiving a 12-lead ECG at the outpatient clinic as standard of care (NOT standard of care)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation detection across 30-second intervals by CardioWatch PPG algorithm vs. 24-48 hour Holter | From enrollment up to 48 hours
  The absolute number of detected AF 30-second intervals by the CardioWatch's PPG algorithm will be determined and compared to the reference ECG holter monitoring, by means of calculating the positive predictive value (PPV), negative predictive value (NPV), specificity, and sensitivity. Performance goals for PPV and NPV are ≥90%, and performance goals for sensitivity and specificity are ≥95%.
Atrial fibrillation detection across 30-second intervals by CardioWatch PPG algorithm vs. short in-clinic 12-lead ECG | From enrollment up to 30 minutes
  The absolute number of detected AF 30-second intervals by the CardioWatch's PPG algorithm will be determined and compared to the reference in-clinic 12-lead ECG, by means of calculating the positive predictive value (PPV), negative predictive value (NPV), specificity, and sensitivity. Performance goals for PPV and NPV are ≥90%, and performance goals for sensitivity and specificity are ≥95%.
Atrial fibrillation detection across 30-second intervals by CardioWatch single-lead ECG vs. 24-48 hour Holter | From enrollment up to 48 hours
  The absolute number of detected AF by the CardioWatch's single-lead ECG algorithm will be determined and compared to the reference ECG holter monitoring at the most similar moment in time by means of calculating the PPV, NPV, specificity, and sensitivity for timestamps corresponding to the single-lead spot checks.
Atrial fibrillation detection across 30-second intervals by CardioWatch single-lead ECG vs. short in-clinic 12-lead ECG | From enrollment up to 30 minutes
  The absolute number of detected AF by the CardioWatch's single-lead ECG algorithm will be determined and compared to the reference in-clinic ECG at the most similar moment in time by means of calculating the PPV, NPV, specificity, and sensitivity for timestamps corresponding to the single-lead spot checks.

SECONDARY OUTCOMES:
Correspondence between cases with AF of greater than 6 minutes, 1 hour, 6 hours, and 12 hours | From enrollment up to 48 hours
  Correspondence between cases with AF of greater than 6 minutes, 1 hour, 6 hours, and 12 hours duration detected by the ECG Holter monitor and the CardioWatch's PPG-algorithm, provided as a percentage of the total cases registered by the ECG Holter monitor for each duration as determined by the Clinical Adjudication Committee (CAC).
Compliance with ECG alerts | From enrollment up to 48 hours
  Compliance with ECG alerts during at home holter-monitoring, together with:
Amount of ECG attempts before successful ECG | From enrollment up to 48 hours
  Amount of ECG attempts before successful ECG during at home holter-monitoring
Confirmation of AF by single-lead ECG | From enrollment up to 48 hours
  The confirmation of AF: single-lead ECG vs PPG-based (ECGs within one hour of alert)
RMSE of HR measurement and reference | From enrollment up to 48 hours
  The root mean square error (RMSE) between the single-lead ECG heart rate (HR) and reference ECG holter HR.
Atrial fibrillation detection performance for males vs. females | Baseline information gathered during enrollment
  Atrial fibrillation detection performance determined for subgroups of males and females individually.
Atrial fibrillation detection performance for BMI subgroups | Baseline information gathered during enrollment
  Atrial fibrillation detection performance determined for subgroups of BMI: Underweight (<18.5); Normal weight (18.5-24.9); Overweight (25-29.9); Obese (≥30).
Atrial fibrillation detection performance for skin colour based subgroups | Baseline information gathered during enrollment
  Atrial fibrillation detection performance determined for subgroups of Skin colour: Monk skin tone (MST) scale 1-3; MST 4-6; MST 7-10. (Researcher will compare reference colors in scale as described in Monk et al. (2023) to the skin of participants)
Atrial fibrillation detection performance for ethinicity based subgroups | Baseline information gathered during enrollment
  Atrial fibrillation detection performance determined for subgroups of Ethnicity: Caucasian; African American; Asian; Hispanic/Latino.
  According to FDA recommendations at least 30 patients total, 15 AF patients and 15 NSR patients, need to be included at each of the subgroup levels of Monk skin tone, ethnicity, sex, BMI. After enrolment of 150 patients, accounting of the subgroups will be considered, and further enrolment will be restricted to ensure minimal distributions of each subgroup level are enrolled, specifically focusing on enrollments in study group D.
Atrial fibrillation detection performance in light of patient activity | From enrollment up to 48 hours
  Atrial fibrillation detection performance for subgroups based on patient activity using ACC: motion; resting; standing
Atrial fibrillation detection performance in light of signal quality index | From enrollment up to 48 hours
  Atrial fibrillation detection performance relative to the signal quality index.

CONTACTS AND LOCATIONS:
Overall Officials: Eelko Ronner, MD, PhD, Principal Investigator — Reinier de Graaf Groep
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No